CLINICAL TRIAL: NCT00206349
Title: Evaluation of Coping Skills in Type 1 Diabetes
Brief Title: Ability to Cope With Type 1 Diabetes
Status: Completed | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Sponsored Programs, Principal Investigator, Baylor College of Medicine
Other Study IDs: 15806
Record Dates: First submitted 2005-09-14; First posted 2005-09-21 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Depression
Keywords: Depression; Socioeconomic status; Type 1 diabetes mellitus; Children; Adolescents
MeSH Terms: conditions — Depression; Diabetes Mellitus, Type 1

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
The purpose of this study is to learn about the relationship that exists between coping skills and blood glucose control. In addition to this, we will study the effect of Type 1 diabetes on coping skills in different age groups, genders, ethnicities, socioeconomic groups, and the duration of diabetes.

DETAILED DESCRIPTION:
Coping with type 1 diabetes can be very difficult. Type 1 diabetes is a very unique chronic disease because it requires constant attention to several responsibilities such as daily glucose monitoring, multiple daily insulin doses, and strict diet and exercise. Several studies have shown that increased rates of poorer glucose control are a result of struggling to cope with type 1 diabetes. This may be due to the fact that many type 1 diabetics experience a feeling of exhaustion, or "burnout," after a certain period of time due to an overwhelming amount of responsibility.

In our study we would like to determine how children's ability to cope with diabetes affects glucose control. By completing several questionnaires, we can analyze different kinds of coping skills through a complex scoring system. These scores will then be analyzed in comparison to your glucose control using HbA1c.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be type 1 diabetic
* English/Spanish speaking
* The legal guardian must be present

Exclusion Criteria:

* Non-cognitive or mentally ill
* Under the age of 8.0 years

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 220
Dates: Start 2004-06; Study Completion 2005-05

CONTACTS AND LOCATIONS:
Overall Officials: Rubina A Heptulla, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States